CLINICAL TRIAL: NCT04238819
Title: A Phase 1b/2 Study of Abemaciclib in Combination With Irinotecan and Temozolomide (Part A) and Abemaciclib in Combination With Temozolomide (Part B) in Pediatric and Young Adult Patients With Relapsed/Refractory Solid Tumors and Abemaciclib in Combination With Dinutuximab, GM-CSF, Irinotecan, and Temozolomide in Pediatric and Young Adult Patients With Relapsed/Refractory Neuroblastoma (Part C)
Brief Title: A Study of Abemaciclib (LY2835219) in Combination With Other Anti-Cancer Treatments in Children and Young Adult Participants With Solid Tumors, Including Neuroblastoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16950; I3Y-MC-JPCS (Other: Eli Lilly and Company); 2019-002931-27 (EudraCT Number); 2023-506778-11-00 (Other: EU Trial Number)
Record Dates: First submitted 2020-01-22; First posted 2020-01-23 (Actual); Results first posted 2025-08-06 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Relapsed Solid Tumor; Refractory Solid Tumor
Keywords: CDK4; CDK6; Ewing's sarcoma; Neuroblastoma; Recurrent neuroblastoma; Malignant rhabdoid tumor; Rhabdomyosarcoma; Osteosarcoma; Brain tumor; Glioblastoma; Malignant glioma; Diffuse intrinsic pontine glioma; Medulloblastoma; Ependymoma; Solid tumor; High-grade glioma
MeSH Terms: conditions — Sarcoma, Ewing; Neuroblastoma; Rhabdoid Tumor; Rhabdomyosarcoma; Osteosarcoma; Brain Neoplasms; Glioblastoma; Glioma; Diffuse Intrinsic Pontine Glioma; Medulloblastoma; Ependymoma | interventions — abemaciclib; Irinotecan; Temozolomide; dinutuximab; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part A Cohort A1 (Experimental): Participants received:
  * Abemaciclib: 70 mg/m², administered orally twice daily (BID).
  * Irinotecan: 50 mg/m²/day, administered IV on Days 1-5 of each cycle.
  * Temozolomide: 100 mg/m²/day, administered orally on Days 1-5 of each cycle.
  Treatment continued until progressive disease, a discontinuation criterion, or unacceptable toxicity. Each cycle lasted 21 days.
  Interventions: Drug: Abemaciclib; Drug: Irinotecan; Drug: Temozolomide
- Part A Cohort A-1 (Experimental): Participants received:
  * Abemaciclib: 55 mg/m², administered orally BID.
  * Irinotecan: 50 mg/m²/day, administered IV on Days 1-5 of each cycle.
  * Temozolomide: 100 mg/m²/day, administered orally on Days 1-5 of each cycle.
  Treatment continued until progressive disease, a discontinuation criterion, or unacceptable toxicity. Each cycle lasted 21 days.
  Interventions: Drug: Abemaciclib; Drug: Irinotecan; Drug: Temozolomide
- Part B Cohort B1 (Experimental): Participants received:
  * Abemaciclib: 70 mg/m², administered orally BID.
  * Temozolomide: 100 mg/m²/day, administered orally on Days 1-5 of each cycle.
  Treatment continued until progressive disease, a discontinuation criterion, or unacceptable toxicity. Each cycle lasted 21 days.
  Interventions: Drug: Abemaciclib; Drug: Temozolomide
- Part B Cohort B2 (Experimental): Participants received:
  * Abemaciclib: 90 mg/m², administered orally BID.
  * Temozolomide: 100 mg/m²/day, administered orally on Days 1-5 of each cycle.
  Treatment continued until progressive disease, a discontinuation criterion, or unacceptable toxicity. Each cycle lasted 21 days.
  Interventions: Drug: Abemaciclib; Drug: Temozolomide
- Part B Cohort B3 (Experimental): Participants received:
  * Abemaciclib: 115 mg/m², administered orally BID.
  * Temozolomide: 100 mg/m²/day, administered orally on Days 1-5 of each cycle.
  Treatment continued until progressive disease, a discontinuation criterion, or unacceptable toxicity. Each cycle lasted 21 days.
  Interventions: Drug: Abemaciclib; Drug: Temozolomide
- Part B Cohort B5 (Experimental): Participants received:
  * Abemaciclib: 115 mg/m², administered orally BID.
  * Temozolomide: 150 mg/m²/day, administered orally on Days 1-5 of each cycle.
  Treatment continued until progressive disease, a discontinuation criterion, or unacceptable toxicity. Each cycle lasted 21 days.
  Interventions: Drug: Abemaciclib; Drug: Temozolomide
- Part C Cohort C1 (Experimental): Participants received:
  * Abemaciclib: 55 mg/m², administered orally BID.
  * Irinotecan: 50 mg/m²/day, administered IV on Days 1-5 of each cycle.
  * Temozolomide: 100 mg/m²/day, administered orally on Days 1-5 of each cycle.
  * Dinutuximab: 17.5mg/m²/day, administered IV on Days 2-5 of each cycle.
  * Granulocyte-macrophage colony-stimulating factor (GM-CSF): 250 μg/m²/day, administered subcutaneously (SC) on Days 6-12 of each cycle.
  Treatment continued until progressive disease, a discontinuation criterion, or unacceptable toxicity. Each cycle lasted 21 days.
  Interventions: Drug: Abemaciclib; Drug: Irinotecan; Drug: Temozolomide; Drug: Dinutuximab; Drug: GM-CSF

INTERVENTIONS:
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219
Drug: Irinotecan — Administered IV
  Arms: Part A Cohort A-1; Part A Cohort A1; Part C Cohort C1
Drug: Temozolomide — Administered orally
Drug: Dinutuximab — Administered IV
  Arms: Part C Cohort C1
Drug: GM-CSF — Administered SC
  Arms: Part C Cohort C1

SUMMARY:
The study's purpose is to see if the drug, abemaciclib, is safe and effective when given with other drugs to kill cancer cells. The study is open to children and young adults with solid tumors, including neuroblastoma, that did not respond or grew during other anti-cancer treatment. For each participant, the study is estimated to last up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Parts A and B only:

  * Participants must be less than or equal to (≤)18 years of age.
  * Body weight greater than or equal to (≥)10 kilograms and body surface area (BSA) ≥0.5
  * Participants with any relapsed/refractory malignant solid tumor (excluding lymphoma), including central nervous system tumors, that have progressed on standard therapies.
  * For sites that are actively enrolling Parts B and C, participants with neuroblastoma who are eligible for Part C will be excluded from Part B unless approved by Lilly CRP/CRS.
* Part C only:

  * Participants must be less than (<) 21 years of age.
  * Participants have a BSA ≥0.2 m².
  * Participants with first relapse/refractory neuroblastoma.
* All Parts

  * Participants must have measurable or evaluable disease by RECIST v1.1 or RANO.
  * A Lansky score ≥50 for participants <16 years of age or Karnofsky score ≥50 for participants ≥16 years of age.
  * Participants must have discontinued all previous treatments for cancer or investigational agents and must have recovered from the acute effects to Grade ≤1 at the time of enrollment.
  * Able to swallow and/or have a gastric/nasogastric tube.
  * Adequate hematologic and organ function ≤2 weeks (14 days) prior to first dose of study drug.
  * Females of reproductive potential must have negative urine or serum pregnancy test at baseline (within 7 days prior to starting treatment).
  * Female participants of reproductive potential must agree to use highly effective contraceptive precautions during the trial. For abemaciclib, females should use contraception for at least 3 weeks following the last abemaciclib. For other study drugs, highly effective contraceptive precautions (and avoiding sperm donation) must be used according to their label.
  * Life expectancy of at least 8 weeks and able to complete at least 1 cycle of treatment.
  * Caregivers and participants willing to make themselves available for the duration of the trial.

Exclusion Criteria:

* Received allogenic bone marrow or solid organ transplant.
* Received live vaccination.
* Intolerability or hypersensitivity to any of the study treatments or its components.
* Diagnosed and/or treated additional malignancy within 3 years prior to enrollment that may affect the interpretation of results, with the exception of curatively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or curatively resected in situ cervical and/or breast cancers.
* Pregnant or breastfeeding.
* Active systemic infections.
* Serious and/or uncontrolled preexisting medical condition(s) that would preclude participation in this study.
* Parts A and C only: Have a bowel obstruction.
* Prior treatment with drugs known to be strong inhibitors or inducers of isoenzyme cytochrome P450 3A (CYP3A) or strong inhibitors of uridine diphosphate-glucuronosyl transferase 1A1 (UGT1A1) if the treatment cannot be discontinued or switched to a different medication at least 5 half-lives prior to starting study drug.
* Received prior treatment with cyclin-dependent kinase (CDK) 4 & 6 inhibitor.
* Part C only: Received prior systemic therapy for relapsed/refractory neuroblastoma.
* Part C only, have received prior anti-GD2 therapy during induction phase.
* Currently enrolled in any other clinical study involving an investigational product or non-approved use of a drug or device.
* Has received an experimental treatment in a clinical trial within the last 30 days or 5 half-lives, whichever is longer.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2025-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (25):
- United States (12):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - The Regents of the University of California - Los Angeles (UCLA Pediatrics), Los Angeles, California
  - Kaiser Permanente Oakland, Oakland, California
  - Kaiser Permanente Roseville, Roseville, California
  - Kaiser Permanente Santa Clara, Santa Clara, California
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - Spectrum Health, Grand Rapids, Michigan
  - Cohen Children's Medical Center, New Hyde Park, New York
  - Atrium Health - Carolinas Medical Center, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania
  - Lifespan Cancer Institute, Providence, Rhode Island
- Perth Children's Hospital, Perth, Western Australia, Australia
- UZ Gent, Ghent, Oost-Vlaanderen, Belgium
- France (3):
  - Centre Leon Berard, Lyon, Rhône
  - Gustave Roussy, Villejuif, Val-de-Marne
  - Institut Curie, Paris
- Germany (3):
  - Universitaetsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitaetsklinikum Essen, Essen, North Rhine-Westphalia
  - Charité Campus Virchow-Klinikum, Berlin
- Fondazione Policlinico Universitario Agostino Gemelli, Rome, Lazio, Italy
- National Cancer Center Hospital, Chuo Ku, Tokyo, Japan
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Hospital Infantil Universitario Niño Jesús, Madrid, Madrid, Comunidad de
  - Hospital Universitari i Politecnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study of Abemaciclib (LY2835219) in Combination With Temozolomide and Irinotecan and Abemaciclib in Combination With Temozolomide in Children and Young Adult Participants With Solid Tumors — https://trials.lillytrialguide.com/en-US/trial/7ojiQLuIsQzitz0DkvlAbe

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A Cohort A1: Participants received:
  * Abemaciclib: 70 milligrams per meters squared (mg/m²), administered orally twice daily (BID).
  * Irinotecan: 50 mg/m²/day, administered intravenously (IV) on Days 1-5 of each cycle.
  * Temozolomide: 100 mg/m²/day, administered orally on Days 1-5 of each cycle. Treatment continued until progressive disease, a discontinuation criterion, or unacceptable toxicity. Each cycle lasted 21 days.
Period: Overall Study
Arm/Group | Part A Cohort A1 | Part A Cohort A-1 | Part B Cohort B1 | Part B Cohort B2 | Part B Cohort B3 | Part B Cohort B5 | Part C Cohort C1
Started | 7 | 13 | 3 | 9 | 3 | 11 | 1
Received At Least One Dose of Study Drug | 7 | 13 | 3 | 9 | 3 | 11 | 1
Completed (A participant was identified as having completed the study if the participant died while on the study or the participant had discontinued study treatment and was in follow up at the time of the final analysis.) | 7 | 13 | 3 | 8 | 2 | 7 | 0
Not Completed | 0 | 0 | 0 | 1 | 1 | 4 | 1
Not completed — Ongoing Treatment | 0 | 0 | 0 | 0 | 1 | 4 | 0
Not completed — Withdrawal by Parent/Subject | 0 | 0 | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A Cohort A1 | Part A Cohort A-1 | Part B Cohort B1 | Part B Cohort B2 | Part B Cohort B3 | Part B Cohort B5 | Part C Cohort C1 | Total
Number analyzed (Participants) | 7 | 13 | 3 | 9 | 3 | 11 | 1 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.9 (3.3) | 12.2 (3.2) | 12.3 (4.7) | 12.2 (4.4) | 9.3 (3.5) | 9.8 (4.5) | 7.00 | 11.4 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 2 | 4 | 3 | 6 | 0 | 23
  Male | 5 | 7 | 1 | 5 | 0 | 5 | 1 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 1 | 2 | 2 | 0 | 7
  Not Hispanic or Latino | 7 | 7 | 2 | 8 | 1 | 9 | 1 | 35
  Unknown or Not Reported | 0 | 4 | 1 | 0 | 0 | 0 | 0 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 3 | 0 | 1 | 0 | 0 | 0 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 7 | 2 | 8 | 3 | 11 | 1 | 36
  More than one race | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  France | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
  Germany | 2 | 1 | 0 | 4 | 0 | 1 | 0 | 8
  Italy | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 3
  Japan | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 5
  Spain | 2 | 7 | 2 | 3 | 3 | 10 | 0 | 27
  United States | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase 2 Dose (RP2D) of Abemaciclib in Combination With Irinotecan and Temozolomide (Part A)
Description: The RP2D of abemaciclib was determined based on the totality of safety, tolerability, and pharmacokinetic results. RP2D of abemaciclib in combination with 50 mg/m²/day irinotecan and 100 mg/m²/day temozolomide on days 1-5 of 21-day cycles was reported.
Time Frame: Cycles 1 and 2 (21 Day Cycles)
Population: All participants in Part A who received at least one dose of abemaciclib and had evaluable data for this outcome.
Measure: Number; unit: milligrams/squared meters (mg/m²) BID
Groups:
- Part A - Abemaciclib: * Cohort A1: 70 mg/m² abemaciclib administered orally BID in combination with 50 mg/m²/day irinotecan administered IV on Days 1-5 of each 21-day cycle and 100 mg/m²/day temozolomide administered orally on Days 1-5 of each 21-day cycle.
  * Cohort A-1: 55 mg/m² abemaciclib administered orally BID in combination with 50 mg/m²/day irinotecan administered IV on Days 1-5 of each 21-day cycle and 100 mg/m²/day temozolomide administered orally on Days 1-5 of each 21-day cycle.
Arm/Group | Part A - Abemaciclib
Number analyzed (Participants) | 20
milligrams/squared meters (mg/m²) BID | 55

2. Primary Outcome: Number or Participants With Dose Limiting Toxicities (DLTs) in Part A
Description: DLT was 1 of the following adverse events likely related to abemaciclib/combination and fulfils any 1 of the following criteria graded per National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0:
  * Any non-hematologic Grade (G) ≥3 toxicity, except:
    * G3 diarrhea lasting <72 hour (h)
    * Acute irinotecan-associated diarrhea lasting <7 days
    * G≥3 nausea, vomiting, constipation that lasts <72 h
    * G3 mucositis/stomatitis lasting <72 h
    * G3 fever/infection
    * G≥3 electrolyte abnormality that lasts <72 h, is not complicated, and resolves spontaneously or responds to conventional medication;
    * G≥3 amylase/lipase that is not associated with symptoms/clinical manifestations of pancreatitis; or
    * AST/ALT elevation resolving to eligibility criteria within 7 days;
  * Hematologic toxicities considered a DLT:
    * A >14-day Cycle 2 delay due to neutropenia/thrombocytopenia
    * G≥3 thrombocytopenia with significant bleeding; or
    * G≥ 4 neutropenic fever
Time Frame: Cycle 1 (21 Day Cycle)
Population: All participants in Part A who received at least one dose of the study drug and had evaluable data for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Cohort A1 | Part A Cohort A-1
Number analyzed (Participants) | 7 | 13
Participants | 3 | 1

3. Primary Outcome: Maximum Tolerated Dose (MTD) of Abemaciclib in Part A
Description: The MTD was defined as the highest dose level at which less than 33% of participants experienced a DLT.
Time Frame: Cycle 1 (21 Days)
Population: All part A participants who received at least one dose of abemaciclib and had evaluable data for this outcome.
Measure: Number; unit: mg/m² BID
Arm/Group | Part A - Abemaciclib
Number analyzed (Participants) | 20
mg/m² BID | 55

4. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time Zero to Tlast (AUC0-tlast) of Abemaciclib in Part A
Description: PK: (AUC0-tlast) was reported.
Time Frame: Pre-dose, 1, 2.5, 4, and 6 hours post Day 1 dose of Cycle 1 and Cycle 2 (21 Day Cycle)
Population: All participants in Part A who received at least one dose of abemaciclib and had evaluable PK data. Per planned analysis, PK analysis was performed as per the dose of study drug received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram *hour per milliliter (ng*h/mL)
Groups:
- Part A: 70 mg/m² Abemaciclib: All part A participants who received 70 mg/m² abemaciclib were included under this arm.
- Part A: 55 mg/m² Abemaciclib: All part A participants who received 55 mg/m² abemaciclib were included under this arm.
Arm/Group | Part A: 70 mg/m² Abemaciclib | Part A: 55 mg/m² Abemaciclib
Number analyzed (Participants) | 6 | 13
nanogram *hour per milliliter (ng*h/mL)
  Cycle 1, Day 1 | 730 (33) | 534 (116)
  Cycle 2, Day 1: number analyzed (Participants) | 2 | 9
  Cycle 2, Day 1 | NA (NA) — Geometric Mean and Geometric Coefficient of Variation couldn't be calculated as there were only two participants. Individual values reported: 373.72 ng*h/mL and 3373.97 ng*h/mL. | 757 (100)

5. Primary Outcome: PK: (AUC0-tlast) of Irinotecan in Part A
Description: PK: AUC0-tlast) was reported.
Time Frame: 2.5, 4, and 6 hours post Day 1 dose of Cycle 1 and Cycle 2 (21 Day Cycle)
Population: All Part A participants who received at least one dose of irinotecan and had evaluable PK data. Per planned analysis, PK analysis was performed as per the dose of drug received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Part A: 50 mg/m²/Day Irinotecan: All part A participants who received 50 mg/m²/day irinotecan were included under this arm.
Arm/Group | Part A: 50 mg/m²/Day Irinotecan
Number analyzed (Participants) | 20
ng*h/mL
  Cycle 1, Day 1 | 1450 (37)
  Cycle 2, Day 1 | 1240 (58)

6. Primary Outcome: PK: (AUC0-tlast) of Temozolomide in Part A
Description: PK: AUC0-tlast was reported.
Time Frame: 1, 2.5, 4, and 6 hours post Day 1 dose of Cycle 1 and Cycle 2 (21 Day Cycle)
Population: All Part A participants who received at least one dose of temozolomide and had evaluable PK data. Per planned analysis, PK analysis was performed as per the dose of drug received.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Part A: 100 mg/m²/Day Temozolomide: All part A participants who received 100 mg/m²/day temozolomide were included under this arm.
Arm/Group | Part A: 100 mg/m²/Day Temozolomide
Number analyzed (Participants) | 19
ng*h/mL
  Cycle 1, Day 1 | 14400 (23)
  Cycle 2, Day 1 | 12200 (44)

7. Primary Outcome: RP2D of Abemaciclib in Combination With Temozolomide (Part B)
Description: The RP2D of abemaciclib was determined based on the totality of safety, tolerability, and pharmacokinetic results. RP2D of abemaciclib in combination with 150 mg/m²/day temozolomide on days 1-5 of 21-day cycles was reported.
Time Frame: Cycles 1 and 2 (21 Day Cycles)
Population: All participants in Part B who received at least one dose of abemaciclib and had evaluable data for this outcome.
Measure: Number; unit: mg/m² BID
Groups:
- Part B - Abemaciclib: Participants received:
  * Abemaciclib: 70 mg/m² or 90 mg/m² or 115 mg/m², administered orally BID.
  * Temozolomide: 100 mg/m²/day or 150 mg/m²/day, administered orally on Days 1-5 of each cycle.
  Treatment continued until progressive disease, a discontinuation criterion, or unacceptable toxicity. Each cycle lasted 21 days.
Arm/Group | Part B - Abemaciclib
Number analyzed (Participants) | 26
mg/m² BID | 115

8. Primary Outcome: Number or Participants With DLTs in Part B
Description: A DLT was 1 of the following adverse events likely related to abemaciclib/combination and fulfils any 1 of the following criteria graded as per National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0:
  * Any non-hematologic Grade (G) ≥3 toxicity, except:
    * G3 diarrhea lasting <72 hr
    * Acute irinotecan-associated diarrhea lasting <7 days
    * G≥3 nausea, vomiting, constipation that lasts <72 hr
    * G3 mucositis/stomatitis lasting <72 hr
    * G3 fever/infection
    * G≥3 electrolyte abnormality that lasts <72 hr, is not complicated, and resolves spontaneously or responds to conventional medication;
    * G≥3 amylase/lipase that is not associated with symptoms/clinical manifestations of pancreatitis; or
    * AST/ALT elevation resolving to eligibility criteria within 7 days;
  * Hematologic toxicities considered a DLT:
    * A >14-day Cycle 2 delay due to neutropenia/thrombocytopenia
    * G≥3 thrombocytopenia with significant bleeding; or
    * G≥ 4 neutropenic fever
Time Frame: Cycle 1 (21 Day Cycle)
Population: All participants in Part B who received at least one dose of the study drug and had evaluable data for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B Cohort B1 | Part B Cohort B2 | Part B Cohort B3 | Part B Cohort B5
Number analyzed (Participants) | 3 | 9 | 3 | 11
Participants | 0 | 1 | 0 | 1

9. Primary Outcome: MTD of Abemaciclib in Part B
Description: The MTD was defined as the highest dose level at which less than 33% of participants experienced a DLT.
Time Frame: Cycle 1 (21 Days)
Population: All participants in Part B who received at least one dose of abemaciclib and had evaluable data for this outcome.
Measure: Number; unit: mg/m² BID
Arm/Group | Part B - Abemaciclib
Number analyzed (Participants) | 26
mg/m² BID | NA — Insufficient number of participants experienced DLT. Thus, MTD could not be calculated.

10. Primary Outcome: PK: AUC0-tlast of Abemaciclib in Part B
Description: PK: AUC0-tlast was reported.
Time Frame: Pre-dose, 1, 2.5, 4, and 6 hours post Day 1 dose of Cycle 1 and Cycle 2 (21 Day Cycle)
Population: All participants in Part B who received at least one dose of abemaciclib and had evaluable PK data. Per planned analysis, PK analysis was performed as per the dose of study drug received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Part B: 70 mg/m² Abemaciclib: All part B participants who received 70 mg/m² abemaciclib were included under this arm.
- Part B: 90 mg/m² Abemaciclib: All part B participants who received 90 mg/m² abemaciclib were included under this arm.
- Part B: 115 mg/m² Abemaciclib: All part B participants who received 115 mg/m² abemaciclib were included under this arm.
Arm/Group | Part B: 70 mg/m² Abemaciclib | Part B: 90 mg/m² Abemaciclib | Part B: 115 mg/m² Abemaciclib
Number analyzed (Participants) | 3 | 8 | 14
ng*h/mL
  Cycle 1, Day 1 | 566 (104) | 728 (60) | 728 (77)
  Cycle 2, Day 1: number analyzed (Participants) | 2 | 5 | 10
  Cycle 2, Day 1 | NA (NA) — Geometric Mean and Geometric Coefficient of Variation couldn't be calculated as there were only two participants. Individual values reported: 994.32 ng*h/mL and 2247.03 ng*h/mL. | 600 (27) | 1060 (57)

11. Primary Outcome: PK: AUC0-tlast of Temozolomide in Part B
Description: PK: AUC0-tlast was reported.
Time Frame: 1, 2.5, 4, and 6 hours post Day 1 dose of Cycle 1 and Cycle 2 (21 Day Cycle)
Population: All Part B participants in who received at least one dose of temozolomide and had evaluable PK data. Per planned analysis, PK analysis was performed as per the dose of drug received.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Part B: 100 mg/m²/Day Temozolomide: All part B participants who received 100 mg/m²/day temozolomide were included under this arm.
- Part B: 150 mg/m²/Day Temozolomide: All part B participants who received 150 mg/m²/day temozolomide were included under this arm.
Arm/Group | Part B: 100 mg/m²/Day Temozolomide | Part B: 150 mg/m²/Day Temozolomide
Number analyzed (Participants) | 13 | 11
ng*h/mL
  Cycle 1, Day 1 | 15800 (19) | 24300 (13)
  Cycle 2, Day 1: number analyzed (Participants) | 13 | 10
  Cycle 2, Day 1 | 15700 (21) | 21100 (43)

12. Primary Outcome: Number of Participants With Overall Response Rate (ORR) in Part C.
Description: ORR: Number of participants with best response of Complete Response (CR), Partial Response (PR), or Minor Response (MR) per International Neuroblastoma Response Criteria (INRC).
  * CR is defined as complete response in all response components:
    * Primary Tumor: <10 mm residual soft tissue primary site and complete resolution of MIBG-avid tumors
    * Soft tissue and bone metastatic response: nonprimary target and nontarget lesions <10 mm and nodes identified as targets decreased to short axis <10mm and MIBG-avid update of nonprimary lesions completely resolved
    * Bone marrow response: no tumor infiltration on reassessment; disappearance of all target lesions;
  * PR is defined as PR in >1component and all other components are either CR, minimal disease (MD) (bone marrow only), PR (soft tissue or bone), or not involved (NI) and no components with progressive disease (PD).
  * MR is defined PR or CR in >1 component and SD in >1 component and no component with PD
Time Frame: Date of first dose to disease progression or death (Up to 25 Months)
Population: All part C participants who received at least one dose of study drug. However, Part C was terminated early and only 1 participant was enrolled in this part.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C Cohort C1
Number analyzed (Participants) | 1
Participants | 1

13. Secondary Outcome: Percentage of Participants With Overall Response Rate (ORR): Part A
Description: ORR: Percentage of participants with best response of CR or PR per Response Evaluation Criteria in Solid Tumors (RECIST) or Response Assessment in Neuro-Oncology (RANO).
  RECIST was used for solid tumors and RANO was used for brain tumors.
  * CR is defined as the disappearance of all target lesions (RECIST) and disappearance of all enhancing measurable and non-measurable disease, no new lesions; stable or improved non-enhancing lesions; and patient must be off corticosteroids and stable or improved clinically (RANO).
  * PR is defined as a 30% decrease in the sum of diameters of target lesions (RECIST) and >50% decrease in the sum of products of perpendicular diameters of all measurable enhancing lesions, no progression of non-measurable disease, no new lesions, stable/improved non-enhancing lesions on same or lower dose of corticosteroids and patient is stable or improved clinically (RANO).
Time Frame: Date of first dose to disease progression or death (Up to 25 Months)
Population: All participants in Part A who received at least one dose of the study drug and had evaluable data for this outcome. Per pre-specified statistical analysis plan, analysis was performed as per the study treatments received.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part A Cohort A1 | Part A Cohort A-1
Number analyzed (Participants) | 7 | 13
Percentage of participants | 0 [NA to NA] — None of the participants achieved ORR. Thus, upper and lower limit of confidence interval values could not be calculated. | 7.7 [0.0 to 22.2]

14. Secondary Outcome: Percentage of Participants With ORR: Part B
Description: as for outcome 13
Time Frame: Date of first dose to disease progression or death (Up to 25 Months)
Population: All participants in Part B who received at least one dose of the study drug and had evaluable data for this outcome. Per pre-specified statistical analysis plan, analysis was performed as per the study treatments received.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part B Cohort B1 | Part B Cohort B2 | Part B Cohort B3 | Part B Cohort B5
Number analyzed (Participants) | 3 | 9 | 3 | 11
Percentage of participants | 0 [NA to NA] — None of the participants achieved ORR. Thus, upper and lower limits of confidence intervals could not be calculated. | 0 [NA to NA] — None of the participants achieved ORR. Thus, upper and lower limits of confidence intervals could not be calculated. | 33.3 [0.0 to 86.7] | 18.2 [0.0 to 41.0]

15. Secondary Outcome: Duration of Response (DoR): Parts A and B.
Description: DoR is the time between first evidence of CR or PR and disease progression or death due to any cause.
  RECIST was used for solid tumors and RANO was used for brain tumors.
  * CR is defined as the disappearance of all target lesions (RECIST) and disappearance of all enhancing measurable and non-measurable disease, no new lesions; stable or improved non-enhancing lesions; and patient must be off corticosteroids and stable or improved clinically (RANO).
  * PR is defined as a 30% decrease in the sum of diameters of target lesions (RECIST) and >50% decrease in the sum of products of perpendicular diameters of all measurable enhancing lesions, no progression of non-measurable disease, no new lesions, stable/improved non-enhancing lesions on same or lower dose of corticosteroids and patient is stable or improved clinically (RANO).
Time Frame: Date of first evidence of a CR or PR to date of objective disease progression or death due to any cause (Up to 25 Months)
Population: All participants in Parts A and B who received at least one dose of the study drug and had evaluable data for this outcome. Per pre-specified statistical analysis plan, analysis was performed as per the study treatments received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part A Cohort A1 | Part A Cohort A-1 | Part B Cohort B1 | Part B Cohort B2 | Part B Cohort B3 | Part B Cohort B5
Number analyzed (Participants) | 0 | 1 | 0 | 0 | 1 | 2
Months |  | 22.59 [NA to NA] — Only 1 participant had events, hence confidence interval limits could not be calculated. |  |  | 7.82 [NA to NA] — Only 1 participant had events, hence confidence interval limits could not be calculated. | 0.03 [NA to NA] — Upper and lower limit confidence intervals cannot be calculated as both participants had the same Duration of Response of 0.03 months.

16. Secondary Outcome: Duration of Response (DoR): Part C
Description: DoR is the time between first evidence of CR, PR or MR and disease progression or death due to any cause.
  CR, PR, and MR was as per International Neuroblastoma Response Criteria (INRC).
  - CR is defined as complete response in all response components: Primary Tumor: <10 mm residual soft tissue primary site and complete resolution of MIBG-avid tumors Soft tissue and bone metastatic response: nonprimary target and nontarget lesions <10 mm and nodes identified as targets decreased to short axis <10mm and MIBG-avid update of nonprimary lesions completely resolved Bone marrow response: no tumor infiltration on reassessment; disappearance of all target lesions;
  * PR is defined as PR in >1 component and all other components are either CR, minimal disease (MD) (bone marrow only), PR (soft tissue or bone), or not involved (NI) and no components with progressive disease (PD).
  * MR is defined PR or CR in >1 component and SD in >1 component and no component with PD
Time Frame: Date of first evidence of a CR, PR, or MR to date of objective disease progression or death due to any cause (Up to 25 Months)
Population: All participants in Part C who received at least one dose of the study drug and had evaluable data for this outcome.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part C Cohort C1
Number analyzed (Participants) | 1
Months | 1.61 [NA to NA] — Only 1 participant had events, hence confidence interval limits could not be calculated.

17. Secondary Outcome: Percentage of Participants With Clinical Benefit Rate (CBR): Part A
Description: The CBR is the percentage of participants with a best response of CR or PR, or Stable Disease (SD) for at least 6 months.
  RECIST was used for solid tumors and RANO was used for brain tumors.
  * CR is defined as the disappearance of all target lesions (RECIST) and disappearance of all enhancing measurable and non-measurable disease, no new lesions; stable or improved non-enhancing lesions; and patient must be off corticosteroids and stable or improved clinically (RANO).
  * PR is defined as a 30% decrease in the sum of diameters of target lesions (RECIST) and >50% decrease in the sum of products of perpendicular diameters of all measurable enhancing lesions, no progression of non-measurable disease, no new lesions, stable/improved non-enhancing lesions on same or lower dose of corticosteroids and patient is stable or improved clinically (RANO).
  * SD is neither sufficient shrinkage nor sufficient increase in the size of the tumor.
Time Frame: Date of first dose to disease progression or death due to any cause (Up to 25 Months)
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part A Cohort A1 | Part A Cohort A-1
Number analyzed (Participants) | 7 | 13
Percentage of participants | 14.3 [0.0 to 40.2] | 30.8 [5.7 to 55.9]

18. Secondary Outcome: Percentage of Participants With CBR: Part B
Description: The CBR is the percentage of participants with a best response of CR or PR, or SD for at least 6 months.
  RECIST was used for solid tumors and RANO was used for brain tumors.
  * CR is defined as the disappearance of all target lesions (RECIST) and disappearance of all enhancing measurable and non-measurable disease, no new lesions; stable or improved non-enhancing lesions; and patient must be off corticosteroids and stable or improved clinically (RANO).
  * PR is defined as a 30% decrease in the sum of diameters of target lesions (RECIST) and >50% decrease in the sum of products of perpendicular diameters of all measurable enhancing lesions, no progression of non-measurable disease, no new lesions, stable/improved non-enhancing lesions on same or lower dose of corticosteroids and patient is stable or improved clinically (RANO).
  * SD is neither sufficient shrinkage nor sufficient increase in the size of the tumor.
Time Frame: Date of first dose to disease progression or death due to any cause (Up to 25 Months)
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part B Cohort B1 | Part B Cohort B2 | Part B Cohort B3 | Part B Cohort B5
Number analyzed (Participants) | 3 | 9 | 3 | 11
Percentage of participants | 33.3 [0.0 to 86.7] | 0 [NA to NA] — None of the participants achieved CBR. Thus, upper and lower limits of confidence intervals could not be calculated. | 33.3 [0.0 to 86.7] | 18.2 [0.0 to 41.0]

19. Secondary Outcome: Percentage of Participants With Disease Control Rate (DCR): Part A
Description: DCR: Percentage of participants with a best overall response of CR, PR, and SD. RECIST was used for solid tumors and RANO was used for brain tumors.
  * CR is defined as the disappearance of all target lesions (RECIST) and disappearance of all enhancing measurable and non-measurable disease, no new lesions; stable or improved non-enhancing lesions; and patient must be off corticosteroids and stable or improved clinically (RANO).
  * PR is defined as a 30% decrease in the sum of diameters of target lesions (RECIST) and >50% decrease in the sum of products of perpendicular diameters of all measurable enhancing lesions, no progression of non-measurable disease, no new lesions, stable/improved non-enhancing lesions on same or lower dose of corticosteroids and patient is stable or improved clinically (RANO).
  * SD is neither sufficient shrinkage nor sufficient increase in the size of the tumor.
Time Frame: Date of first dose to measured progressive disease (Up to 25 Months)
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part A Cohort A1 | Part A Cohort A-1
Number analyzed (Participants) | 7 | 13
Percentage of participants | 71.4 [38.0 to 100.0] | 53.8 [26.7 to 80.9]

20. Secondary Outcome: Percentage of Participants With DCR: Part B
Description: as for outcome 19
Time Frame: Date of first dose to measured progressive disease (Up to 25 Months)
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part B Cohort B1 | Part B Cohort B2 | Part B Cohort B3 | Part B Cohort B5
Number analyzed (Participants) | 3 | 9 | 3 | 11
Percentage of participants | 33.3 [0.0 to 86.7] | 55.6 [23.1 to 88.0] | 100 [100.0 to 100.0] | 36.4 [7.9 to 64.8]

21. Secondary Outcome: Progression-Free Survival (PFS): Part C
Description: Progression-free survival is measured as the time from first dose of study drug to progressive disease or death, whichever occurs first. PFS for Part C was reported.
Time Frame: Date of first dose to progressive disease or death (Up to 25 Months)
Population: as for outcome 12
Measure: Number; unit: Months
Arm/Group | Part C Cohort C1
Number analyzed (Participants) | 1
Months | 2.9

22. Secondary Outcome: Abemaciclib Tablet Acceptability
Description: Participants were evaluated for abemaciclib acceptability (palatability and ease of administration) by asking a question - " Was it easy or difficult for the study subject to swallow the abemaciclib today?" Participants or their caregivers or both could respond using the following possible answers: Very difficult, difficult, neither easy nor difficult, easy, or very easy.
Time Frame: Cycle 1 Day 1, Cycle 1 Day 15, and Cycle 2 Day 1 (21 Day Cycles)
Population: All participants in Parts A and B, who received at least one dose of abemaciclib and had evaluable data for this outcome. Per protocol, data were summarized by responses provided by participants, and/or caregivers on the acceptability of the abemaciclib received on Cycle 1 Day 1, Cycle 1 Day 15, and Cycle 2 Day 1.
Measure: Count of Participants; unit: Participants
Groups:
- Part A Cohort A1 (Caregiver Responses - Cycle 1 Day 1); Part A Cohort A1 (Caregiver Responses - Cycle 1 Day 15); Part A Cohort A1 (Caregiver Responses - Cycle 2 Day 1); Part A Cohort A1 (Participant Responses - Cycle 1 Day 1); Part A Cohort A1 (Participant Responses - Cycle 1 Day 15); Part A Cohort A1 (Participant Responses - Cycle 2 Day 1): Participants received:
  * Abemaciclib: 70 milligrams per meters squared (mg/m²), administered orally twice daily (BID).
  * Irinotecan: 50 mg/m²/day, administered intravenously (IV) on Days 1-5 of each cycle.
  * Temozolomide: 100 mg/m²/day, administered orally on Days 1-5 of each cycle.
  Treatment continued until progressive disease, a discontinuation criterion, or unacceptable toxicity. Each cycle lasted 21 days.
- Part A Cohort A-1(Caregiver Responses - Cycle 1 Day 1); Part A Cohort A-1(Caregiver Responses - Cycle 1 Day 15); Part A Cohort A-1(Caregiver Responses - Cycle 2 Day 1); Part A Cohort A-1(Participant Responses - Cycle 1 Day 1); Part A Cohort A-1(Participant Responses - Cycle 1 Day 15); Part A Cohort A-1(Participant Responses - Cycle 2 Day 1): Participants received:
  * Abemaciclib: 55 mg/m², administered orally BID.
  * Irinotecan: 50 mg/m²/day, administered IV on Days 1-5 of each cycle.
  * Temozolomide: 100 mg/m²/day, administered orally on Days 1-5 of each cycle.
  Treatment continued until progressive disease, a discontinuation criterion, or unacceptable toxicity. Each cycle lasted 21 days.
- Part B Cohort B1 (Caregiver Responses - Cycle 1 Day 1); Part B Cohort B1 (Caregiver Responses - Cycle 1 Day 15); Part B Cohort B1 (Caregiver Responses - Cycle 2 Day 1); Part B Cohort B1 (Participant Responses - Cycle 1 Day 1); Part B Cohort B1 (Participant Responses - Cycle 1 Day 15); Part B Cohort B1 (Participant Responses - Cycle 2 Day 1): Participants received:
  * Abemaciclib: 70 mg/m², administered orally BID.
  * Temozolomide: 100 mg/m²/day, administered orally on Days 1-5 of each cycle.
  Treatment continued until progressive disease, a discontinuation criterion, or unacceptable toxicity. Each cycle lasted 21 days.
- Part B Cohort B2 (Caregiver Responses - Cycle 1 Day 1); Part B Cohort B2 (Caregiver Responses - Cycle 1 Day 15); Part B Cohort B2 (Caregiver Responses - Cycle 2 Day 1); Part B Cohort B2 (Participant Responses - Cycle 1 Day 1); Part B Cohort B2 (Participant Responses - Cycle 1 Day 15); Part B Cohort B2 (Participant Responses - Cycle 2 Day 1): Participants received:
  * Abemaciclib: 90 mg/m², administered orally BID.
  * Temozolomide: 100 mg/m²/day, administered orally on Days 1-5 of each cycle.
  Treatment continued until progressive disease, a discontinuation criterion, or unacceptable toxicity. Each cycle lasted 21 days.
- Part B Cohort B3 (Caregiver Responses - Cycle 1 Day 1); Part B Cohort B3 (Caregiver Responses - Cycle 1 Day 15); Part B Cohort B3 (Caregiver Responses - Cycle 2 Day 1); Part B Cohort B3 (Participant Responses - Cycle 1 Day 1); Part B Cohort B3 (Participant Responses - Cycle 1 Day 15); Part B Cohort B3 (Participant Responses - Cycle 2 Day 1): Participants received:
  * Abemaciclib: 115 mg/m², administered orally BID.
  * Temozolomide: 100 mg/m²/day, administered orally on Days 1-5 of each cycle.
  Treatment continued until progressive disease, a discontinuation criterion, or unacceptable toxicity. Each cycle lasted 21 days.
- Part B Cohort B5 (Caregiver Responses - Cycle 1 Day 1); Part B Cohort B5 (Caregiver Responses - Cycle 1 Day 15); Part B Cohort B5 (Caregiver Responses - Cycle 2 Day 1); Part B Cohort B5 (Participant Responses - Cycle 1 Day 1); Part B Cohort B5 (Participant Responses - Cycle 1 Day 15); Part B Cohort B5 (Participant Responses - Cycle 2 Day 1): Participants received:
  * Abemaciclib: 115 mg/m², administered orally BID.
  * Temozolomide: 150 mg/m²/day, administered orally on Days 1-5 of each cycle.
  Treatment continued until progressive disease, a discontinuation criterion, or unacceptable toxicity. Each cycle lasted 21 days.
Arm/Group | Part A Cohort A1 (Caregiver Responses - Cycle 1 Day 1) | Part A Cohort A1 (Caregiver Responses - Cycle 1 Day 15) | Part A Cohort A1 (Caregiver Responses - Cycle 2 Day 1) | Part A Cohort A1 (Participant Responses - Cycle 1 Day 1) | Part A Cohort A1 (Participant Responses - Cycle 1 Day 15) | Part A Cohort A1 (Participant Responses - Cycle 2 Day 1) | Part A Cohort A-1(Caregiver Responses - Cycle 1 Day 1) | Part A Cohort A-1(Caregiver Responses - Cycle 1 Day 15) | Part A Cohort A-1(Caregiver Responses - Cycle 2 Day 1) | Part A Cohort A-1(Participant Responses - Cycle 1 Day 1) | Part A Cohort A-1(Participant Responses - Cycle 1 Day 15) | Part A Cohort A-1(Participant Responses - Cycle 2 Day 1) | Part B Cohort B1 (Caregiver Responses - Cycle 1 Day 1) | Part B Cohort B1 (Caregiver Responses - Cycle 1 Day 15) | Part B Cohort B1 (Caregiver Responses - Cycle 2 Day 1) | Part B Cohort B1 (Participant Responses - Cycle 1 Day 1) | Part B Cohort B1 (Participant Responses - Cycle 1 Day 15) | Part B Cohort B1 (Participant Responses - Cycle 2 Day 1) | Part B Cohort B2 (Caregiver Responses - Cycle 1 Day 1) | Part B Cohort B2 (Caregiver Responses - Cycle 1 Day 15) | Part B Cohort B2 (Caregiver Responses - Cycle 2 Day 1) | Part B Cohort B2 (Participant Responses - Cycle 1 Day 1) | Part B Cohort B2 (Participant Responses - Cycle 1 Day 15) | Part B Cohort B2 (Participant Responses - Cycle 2 Day 1) | Part B Cohort B3 (Caregiver Responses - Cycle 1 Day 1) | Part B Cohort B3 (Caregiver Responses - Cycle 1 Day 15) | Part B Cohort B3 (Caregiver Responses - Cycle 2 Day 1) | Part B Cohort B3 (Participant Responses - Cycle 1 Day 1) | Part B Cohort B3 (Participant Responses - Cycle 1 Day 15) | Part B Cohort B3 (Participant Responses - Cycle 2 Day 1) | Part B Cohort B5 (Caregiver Responses - Cycle 1 Day 1) | Part B Cohort B5 (Caregiver Responses - Cycle 1 Day 15) | Part B Cohort B5 (Caregiver Responses - Cycle 2 Day 1) | Part B Cohort B5 (Participant Responses - Cycle 1 Day 1) | Part B Cohort B5 (Participant Responses - Cycle 1 Day 15) | Part B Cohort B5 (Participant Responses - Cycle 2 Day 1)
Number analyzed (Participants) | 3 | 2 | 5 | 7 | 5 | 6 | 6 | 4 | 7 | 10 | 8 | 8 | 2 | 1 | 1 | 2 | 1 | 2 | 5 | 4 | 4 | 6 | 6 | 6 | 1 | 1 | 1 | 3 | 3 | 3 | 6 | 7 | 4 | 9 | 9 | 9
Participants
  Very easy to swallow tablet | 1 | 1 | 3 | 4 | 4 | 4 | 6 | 4 | 6 | 6 | 4 | 5 | 1 | 0 | 0 | 2 | 1 | 2 | 3 | 3 | 2 | 5 | 5 | 3 | 0 | 1 | 1 | 3 | 3 | 3 | 3 | 6 | 4 | 6 | 8 | 9
  Easy to swallow tablet | 2 | 1 | 2 | 3 | 1 | 2 | 0 | 0 | 1 | 4 | 3 | 3 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
  Neither easy nor difficult to swallow tablet | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0
  Difficult to swallow tablet | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Very difficult to swallow tablet | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline Up To 112 Weeks
Description: All participants who received at least one dose of the study drug. Gender specific events occurring only in male or female participants have had the number of participants at risk adjusted accordingly. The adverse events were analyzed and reported according to the study treatments pre-specified in the protocol.
Groups:
- Part A Cohort A1: Participants received:
  * Abemaciclib: 70 mg/m², administered orally BID.
  * Irinotecan: 50 mg/m²/day, administered IV on Days 1-5 of each cycle.
  * Temozolomide: 100 mg/m²/day, administered orally on Days 1-5 of each cycle.
  Treatment continued until progressive disease, a discontinuation criterion, or unacceptable toxicity. Each cycle lasted 21 days.
- Part C Cohort C1: Participants received:
  * Abemaciclib: 55 mg/m², administered orally BID.
  * Irinotecan: 50 mg/m²/day, administered IV on Days 1-5 of each cycle.
  * Temozolomide: 100 mg/m²/day, administered orally on Days 1-5 of each cycle.
  * Dinutuximab: 17.5mg/m²/day, administered IV on Days 2-5 of each cycle.
  * GM-CSF: 250 μg/m²/day, administered SC on Days 6-12 of each cycle.
  Treatment continued until progressive disease, a discontinuation criterion, or unacceptable toxicity. Each cycle lasted 21 days.
Arm/Group | Part A Cohort A1 | Part A Cohort A-1 | Part B Cohort B1 | Part B Cohort B2 | Part B Cohort B3 | Part B Cohort B5 | Part C Cohort C1
All-Cause Mortality (participants affected / at risk) | 1/7 | 1/13 | 0/3 | 1/9 | 1/3 | 1/11 | 0/1
Serious Adverse Events (participants affected / at risk) | 3/7 | 5/13 | 2/3 | 0/9 | 0/3 | 3/11 | 1/1
Other Adverse Events (participants affected / at risk) | 7/7 | 13/13 | 3/3 | 8/9 | 3/3 | 11/11 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Cohort A1 (N=7) | Part A Cohort A-1 (N=13) | Part B Cohort B1 (N=3) | Part B Cohort B2 (N=9) | Part B Cohort B3 (N=3) | Part B Cohort B5 (N=11) | Part C Cohort C1 (N=1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vancomycin infusion reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part A Cohort A1 (N=7) | Part A Cohort A-1 (N=13) | Part B Cohort B1 (N=3) | Part B Cohort B2 (N=9) | Part B Cohort B3 (N=3) | Part B Cohort B5 (N=11) | Part C Cohort C1 (N=1)
Anaemia (Blood and lymphatic system disorders) | 5 (11) | 8 (17) | 1 (1) | 5 (5) | 1 (2) | 7 (9) | 1 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 6 (16) | 4 (21) | 1 (1) | 2 (9) | 2 (3) | 8 (13) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 4 (4) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 6 (25) | 10 (35) | 2 (3) | 6 (17) | 3 (10) | 8 (20) | 1 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (15) | 8 (29) | 2 (2) | 4 (8) | 2 (7) | 9 (16) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0/5 (0) | 1/7 (1) | 0/1 (0) | 0/5 (0) | 0 (0) | 0/5 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cushing's syndrome (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anisocoria (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blepharospasm (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema eyelids (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ophthalmoplegia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 4 (10) | 6 (11) | 1 (1) | 2 (2) | 2 (7) | 4 (7) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal pruritus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal rash (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (9) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (18) | 13 (65) | 0 (0) | 5 (22) | 3 (6) | 9 (24) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (17) | 5 (13) | 0 (0) | 2 (4) | 1 (1) | 4 (4) | 1 (9)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue atrophy (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (18) | 7 (21) | 1 (1) | 6 (12) | 2 (3) | 5 (10) | 1 (9)
Catheter site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (3) | 5 (6) | 1 (2) | 2 (3) | 0 (0) | 2 (5) | 1 (2)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Pyrexia (General disorders) | 1 (3) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 3 (5) | 1 (7)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial diarrhoea (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis cryptosporidial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes dermatitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superinfection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 4 (13) | 4 (9) | 1 (2) | 1 (1) | 1 (1) | 2 (3) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 4 (10) | 3 (6) | 0 (0) | 0 (0) | 1 (2) | 3 (6) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 2 (5) | 1 (2) | 0 (0) | 2 (5) | 2 (4) | 5 (10) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystatin c increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (3) | 1 (2) | 1 (1) | 1 (2) | 1 (1) | 3 (3) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 3 (3) | 6 (19) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 5 (9) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 1 (6) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (4) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3) | 3 (7) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 2 (5) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Vitamin b12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (5) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anterograde amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotonia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paresis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device malfunction (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital rash (Reproductive system and breast disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0/5 (0) | 0/7 (0) | 0/1 (0) | 0/5 (0) | 0 (0) | 1/5 (1) | 0 (0)
Vulvovaginal inflammation (Reproductive system and breast disorders) | 0/2 (0) | 0/6 (0) | 0/2 (0) | 0/4 (0) | 0 (0) | 1/6 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (3)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-07-18): https://cdn.clinicaltrials.gov/large-docs/19/NCT04238819/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/19/NCT04238819/SAP_001.pdf